CLINICAL TRIAL: NCT00159991
Title: Arterial Revascularization for Coronary Bypass Surgery: A Randomized Trial Comparing the Outcome After Using LIMA + Vein Grafts Versus Total Arterial Revascularization With LIMA + RIMA + Radial Artery Grafts
Brief Title: Copenhagen Arterial Revascularization Randomized Patency and Outcome Trial
Acronym: CARRPO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Heart Foundation (Other); Lundbeck Foundation (Other); Copenhagen Hospital Corporation (Other)
Responsible Party: Sune Damgaard MD, Department of Cardiothoracic Surgery, Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 961502837
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Arteriosclerosis; Ischemic Heart Disease; Angina Pectoris
Keywords: Coronary artery bypass grafting; Total arterial revascularization; Internal mammary artery grafting; Radial artery grafting
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Angina Pectoris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Total arterial revascularization
  Interventions: Procedure: Total arterial revascularization
- B (Active Comparator): Conventional revascularization
  Interventions: Procedure: Conventional revascularization

INTERVENTIONS:
Procedure: Total arterial revascularization — Coronary artery bypass grafting using LIMA and RIMA and/or radial artery grafts
  Other Names: LIMA: left internal mammary artery; RIMA: right internal mammary artery
  Arms: A
Procedure: Conventional revascularization — Coronary artery bypass grafting using LIMA and saphenous vein grafts
  Other Names: LIMA: left internal mammary artery
  Arms: B

SUMMARY:
There is a remarkable lack of randomized trials concerning the potential benefit of using arterial conduits for coronary bypass surgery. This is the purpose of the present trial. Exclusive use of arterial conduits might result in improved conduit viability, reduced risk of recurrent angina, myocardial infarction and other cardiac events, reduced need for antianginal medication, improved functional status and possibly improved long term survival. The patients will be followed for ten years after surgery.

DETAILED DESCRIPTION:
I: Background

There is a remarkable lack of randomized studies concerning the potential benefit of using arterial grafts for coronary revascularization. Numerous observational reports consistently confirm, that the use of a LIMA-LAD grafts is not associated with increased peroperative mortality or morbidity and will result in an approximately 10% improved survival at 10 years postoperatively.

The average patency for LIMA-LAD grafts is 80%-85% after 10 years. 50% of the vein grafts are occluded. LIMA-LAD grafting reduces the risk of of late myocardial infarction, other cardiac events and reoperation, however the effect on recurrent angina or need of antianginal medication is less certain.

The question, whether bilateral IMA grafting has long term benefits compared to single IMA grafts is controversial. Numerous observational retrospective studies fail to demonstrate convincingly, that bilateral IMA grafting reduces long term mortality and improves the frequency of late cardiac events and recurrent angina, but these data are difficult to compare due to selection bias. It is not quite clear, if a minimal benefit represents a true difference in outcome, or if two different populations are compared.

Whether an increased degree of arterial revascularization, including radial artery (RA) and IMA grafts, will result in an improved long term survival, reduced risk for recurrent angina, reinfarction, antianginal medication and improved quality of life, is unclear.

A randomized trial has not yet been performed and current observational 5 year follow-up data are promising, but cannot document an anticipated benefit from a more stringent scientific point of view.

II: Hypothesis

Coronary bypass grafting with the use of LIMA + RIMA + RA (total arterial revascularization) vs. LIMA + saphenous vein grafts will result in equal peroperative mortality and morbidity rates and improve long term outcome in terms of improved patency rates, reduced risk of recurrent angina, infarction and other cardiac events, reduced need for antianginal medication, improved functional status and possibly improved long term survival.

III: Aim of the study

Prospective randomized trial comparing coronary bypass grafting with the use of LIMA + RIMA + RA vs. LIMA + saphenous vein grafts in patients with 2 or 3 vessel disease (more than 1 graft anticipated) with respect to:

1. Graft patency rates at 1, 5 and 10 years postoperatively
2. Cardiac event free survival 1, 5 and 10 years postoperatively (risk of hospital readmission due to infarction, suspicion of infarction, unstable angina, arrythmias, heart insufficiency, need for renewed angiography, angioplasty, redo surgery)
3. Peroperative mortality and morbidity
4. Risk of recurrent angina and need for antianginal medication 1, 5 and 10 years postoperatively
5. Data on functional status and social rehabilitation at clinical controls 3 months, 1, 5 and 10 years postoperatively

IV: Design & methods

1. Design

   Prospective randomized trial. Patients will be randomized into 2 groups:

   Group A: Arterial revascularization with LIMA + RIMA + RA.

   Group B: LIMA and saphenous vein grafts are used as graft material.
2. Inclusion criteria

   * Patients with 2 or 3 vessel coronary artery disease, where more than 1 coronary bypass graft is anticipated.
   * Elective or subacute operation (unstable AP with surgery within a few days)
   * Inclusion is independent of ventricular function, recent MI, degree and type of coronary lesions and secondary risk factors as diabetes, hyperlipidemia, hypertension, lung function, chronic obstructive lung disease, peripheral atherosclerotic disease, kidney function, earlier cerebrovascular disease.
   * Age: < 70 years.
   * Sufficient collateral blood supply to the hand by the ulnar artery, evaluated by the Allen test.
   * Patients must be able to give informed consent.
3. Exclusion criteria

   * Concurrent malignant disease with expected survival of < 5 years.
   * Unsuitable saphenous vein grafts evaluated preoperatively.
   * Unsuitable saphenous vein grafts with a diameter > 6mm evaluated peroperatively.
   * Acute operation (unstable hemodynamics in terms of need of inotropic support, ongoing MI with dynamic ECG changes, cardiogenic shock).
   * Concommitant operation for valve disease or other forms of heart surgery.
   * Redo operations.
4. Surgery, anaesthesia and postoperative care

   Surgery, anaesthesia and postoperative care are performed according to current guidelines at our institution.
5. Endpoints and follow-up

   The study is designed with respect to two primary endpoints:
   1. Distal anastomotic patency rates at 1, 5 and 10 years postoperatively
   2. Cardiac event free survival 1, 5 and 10 years postoperatively (Cardiac event free survival is defined as survival without readmission due to infarction, suspicion of infarction, unstable angina, arrythmias, heart insufficiency, need for renewed angiography, angioplasty, redo surgery)

   Secondary endpoints:
   1. Peroperative mortality and morbidity (frequency of peroperative/ postoperative infarction, arrythmias, use of IABP, inotropic support, pulmonary, renal and cerebral complications, length of stay in the ICU, etc. according to registration schemes).
   2. Risk of recurrent angina and need for antianginal medication 1, 5 and 10 years postoperatively
   3. Data on functional status and social rehabilitation at clinical controls 3 months, 1, 5 and 10 years postoperatively

   According to these endpoints the follow-up is planned as:
   * 3 month clinical control at referring hospitals
   * 1 year control including angiography, which can be performed on an outpatient basis.
   * 5 year control including conventional angiography and computed tomography angiography.
   * 10 year control including computed tomography angiography, which can be performed on an outpatient basis.
6. Statistics

Sample size is calculated with respect to the primary endpoint graft patency at 1 and 5 years. A difference of 10-15% of patency in favour of the radial artery as bypass graft is regarded as clinically relevant. Observational data on radial artery patency indicate patency rates of 90-95% at 1 year and 85% at 5 years, while saphenous vein graft patency is 80-90% at 1 year and 60-70% at 5 years.

To detect such a difference (15% improved patency for RA grafts, 85% vs 70%) with a 90% probability (type 2 error 0.10) and a significance level of 0.05, the sample size for each group would be n=150.

A 15% difference in patency rates at 5 years is in our opinion an assumption that probably overestimates the vein graft patency, which means, that a sample size of 150 patients in each group should guarantee with a high probability a statistically significant outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 2 or 3 vessel coronary artery disease, where more than 1 coronary bypass graft is anticipated.
* Elective or subacute operation (unstable AP with surgery within a few days)
* Inclusion is independent of ventricular function, recent MI, degree and type of coronary lesions and secondary risk factors as diabetes, hyperlipidemia, hypertension, lung function, chronic obstructive lung disease, peripheral atherosclerotic disease, kidney function, earlier cerebrovascular disease.
* Age: < 70 years.
* Sufficient collateral blood supply to the hand by the ulnar artery, evaluated by the Allen test.
* Patients must be able to give informed consent.

Exclusion Criteria:

* Concurrent malignant disease with expected survival of < 5 years.
* Unsuitable saphenous vein grafts evaluated preoperatively.
* Unsuitable saphenous vein grafts with a diameter > 6mm evaluated preoperatively.
* Acute operation (unstable hemodynamics in terms of need of inotropic support, ongoing MI with dynamic ECG changes, cardiogenic shock).
* Concommitant operation for valve disease or other forms of heart surgery. Redo operations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2002-02; Primary Completion 2011-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Angiographic distal anastomotic patency rates | 1, 5 and 10 years postoperatively
Cardiac event free survival | 1, 5 and 10 years postoperatively

SECONDARY OUTCOMES:
Peroperative mortality | Until 3 months postoperatively
Postoperative morbidity (frequency of peroperative/ postoperative infarction, arrythmias, use of IABP, inotropic support, pulmonary, renal and cerebral complications, length of stay in the ICU, etc. according to registration schemes). | 3 months postoperatively
Risk of recurrent angina and need for antianginal medication | 1, 5 and 10 years postoperatively
Data on functional status and social rehabilitation at clinical controls | 3 months, 1, 5 and 10 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Sune Damgaard, MD, Principal Investigator — Dept. of Cardiothoracic Surgery, Rigshospitalet, Copenhagen; Daniel A Steinbrüchel, Professor, Study Director — Dept. of Cardiothoracic Surgery, Rigshospitalet, Copenhagen; Jens T Lund, Consultant, Study Chair — Dept. of Cardiothoracic Surgery, Rigshospitalet, Copenhagen; Henning Kelbæk, Consultant, Study Chair — Cardiac Cath. Lab., Rigshospitalet, Copenhagen; Jan K Madsen, Consultant, Study Chair — Dept. of Cardiology, Gentofte County Hospital, Copenhagen
Locations (1):
- Department of Cardiothoracic Surgery, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Damgaard S, Wetterslev J, Lund JT, Lilleor NB, Perko MJ, Kelbaek H, Madsen JK, Steinbruchel DA. One-year results of total arterial revascularization vs. conventional coronary surgery: CARRPO trial. Eur Heart J. 2009 Apr;30(8):1005-11. doi: 10.1093/eurheartj/ehp048. Epub 2009 Mar 6. PMID 19270315